CLINICAL TRIAL: NCT01842074
Title: Desensitization With Bortezomib Before a Living Kidney Donation
Acronym: VELDON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110147; 2012-001988-78 (EudraCT Number)
Record Dates: First submitted 2013-04-08; First posted 2013-04-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Patients Awaiting a Living Kidney Donation
Keywords: bortezomib; desensitization; living kidney transplantation
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): Pilot study on the efficacy and safety of bortezomib during desensitization before a living kidney donation
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Pilot study on the efficacy and safety of bortezomib during desensitization before a living kidney donation

SUMMARY:
The investigators plan to study the role of bortezomib for desensitizing patients awaiting a living kidney donation who have a titer of Donor Specific anti human leucocyte antigen (HLA) Antibody (DSA) between 1000 and 3000 MFI with a pilot study of 10 patients recruited in 4 hospital in FRANCE.

DETAILED DESCRIPTION:
The investigators plan to study the role of bortezomib for desensitizing patients awaiting a living kidney donation who have a titer of Donor Specific anti HLA Antibody (DSA) between 1000 and 3000 MFI with a multicentre pilot study of 10 patients. The effect of bortezomib will be observed up to 6 month after bortezomib treatment prior to transplantation and 12 month after transplantation if performed. The living kidney donation will be performed only if the DSA level drops below 1000 MFI which means an efficacy of the desensitization.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 70 years old
* awaiting a living kidney donation
* but with a least one DSA titer between 1000 MFI and 3000 MFI

Exclusion Criteria:

* positive cell dependent cytotoxicity CM,
* DSA level above 3000 MFI
* and every condition that is a contre indication for bortezomib treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Donor specific antibody (DSA) level below 1000MFI authorizing the living kidney donation | up 6 months after bortezomib treatment and before transplantation
  Bortezomib treatment should allow a decrease in DSA level below a threshold level authorizing the living kidney donation with minimal risk

SECONDARY OUTCOMES:
Absolute and relative differences of the DSA titer ans antiHLA non DSA titer bortezomib treatment | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment 12 months after transplantation if performed, if not 6 month after the last bortezomib injection
Frequency of clinical symptoms and anomalies | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment
Frequency of side effects | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment
Frequency of anomalies at the standard blood tests | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment
Frequency of anomalies at the total lymphocyte count and phenotyping | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment
Frequency of proteinuria and anomalies at the glomerular filtration rate | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment
Proportion of transplanted patients | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment 12 months after transplantation if performed, if not 6 month after the last bortezomib injection
Incidence of biopsy proven acute rejection and chronic rejection | 12 month after the living kidney donation if performed or 6 month after the last bortezomib injection if the living kidney donation could not be performed
  Safety and efficacy of bortezomib treatment 12 months after transplantation if performed, if not 6 month after the last bortezomib injection

CONTACTS AND LOCATIONS:
Overall Officials: Hélène François, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris - Bicêtre Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Bicêtre Hospital, Le Kremlin-Bicêtre, France